CLINICAL TRIAL: NCT05140395
Title: Clinical Perfomance Study of the ABTEST© Card in Vitro Medical Device
Brief Title: ABTEST© Card Clinical Perfomance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diagast (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPSP_20-01_V1
Record Dates: First submitted 2021-11-19; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Transfusion Reaction
Keywords: Reagent Kits, Diagnostic
MeSH Terms: conditions — Transfusion Reaction; Disease

STUDY DESIGN:
Intervention Model Description: in situ used for near patient In vitro Medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre transfusion control (Experimental): Pre control transfusion with the referent reagent and the in study reagent
  Interventions: Diagnostic Test: ABTEST card

INTERVENTIONS:
Diagnostic Test: ABTEST card — Pre transfusional control with the referent ABTEST card and the in study ABDTEST Card

SUMMARY:
The study confirms the performance equivalence of the in vitro Diagnostic reagent ABTEST card used with the new reformulated WS solution

DETAILED DESCRIPTION:
The study consists to perform on 100 patients a first pre transfusional control with the reference in vitro reagent ABTEST card (CE Marked reagent) followed by a another pre transfusional control with the in vitro reagent ABTEST card in study (new reformulated WS solution used) .

ELIGIBILITY:
66 patients in hematology / oncology departments , including 20 patients with a hemoglobin significantly below the norm (<8g / dl hemoglobin in the blood), and about to receive a transfusion. 20 patients hospitalized in gastroenterology with a transfusion need 4 internal medicine patients with cold agglutinins, in a transfusion context or not.

10 neonatal patients, background transfusion or Guthrie test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Agreement between two reagents | 5 minutes
  performance of pre transfusional controls with the referent reagent and the reagent in study

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Huchette, phD, Principal Investigator — CH Arras
Locations (1):
- CH Arras, Arras, France

IPD SHARING:
Plan to Share IPD: No